CLINICAL TRIAL: NCT02598531
Title: Surgical Weight-Loss to Improve Functional Status Trajectories Following Total Knee Arthroplasty (SWIFT Trial)
Acronym: SWIFT
Status: Terminated | Type: Observational
Why Stopped: Recruitment Failure
Sponsor: Geisinger Clinic (Other)
Collaborators: NYU Langone Health (Other); University of Virginia (Other); State University of New York at Buffalo (Other); University of Rochester (Other); Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0244
Record Dates: First submitted 2015-10-23; First posted 2015-11-06 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Osteoarthritis
MeSH Terms: conditions — Obesity; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples Synovial Fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test Arm: Test Arm participants will be enrolled in the standard of care bariatric surgery program and will undergo surgical weight loss through Laparoscopic Sleeve Gastrectomy or Laparoscopic Gastric Bypass. Approximately 9-13 months post surgery, each participant will be evaluated to determine if he/she is still eligible for a total knee replacement or if their need has been removed. If still eligible, participants will be enrolled in the standard of care TKA program and will undergo a TKA procedure. Participants will complete nine (9) research visits over 3.5-4 years.
- Control Arm: Control Arm participants will be enrolled in the standard of care TKA program and complete six (6) research visits over 2.5-3 years. This group of participants will undergo a TKA procedure without any surgical weight loss intervention.

SUMMARY:
The purpose of the SWIFT Trial is to answer two research questions.

1. Does bariatric surgery before total knee arthroplasty (TKA) improve both perioperative and long-term outcomes of TKA in extreme obesity?
2. Does bariatric surgery before TKA delay or possibly negate the need for arthroplasty?

DETAILED DESCRIPTION:
Obese patients pursing a TKA procedure are typically encouraged to lose weight prior to the procedure as part of the patient's treatment plan. If the patient chooses to receive treatment for his or her obesity, the Orthopedic provider may refer the patient to a weight management provider. If a patient is eligible for TKA and meets the inclusion and exclusion criteria (containing BMI and corresponding comorbidity measures), he/she is eligible to participate in the study.

In this study there will be two arms, a Test Arm in which patients undergo bariatric surgery prior to TKA and a Control Arm in which patients undergo TKA only. Patients will choose which arm they enter, based on whether or not they want to undergo surgical weight loss intervention prior to TKA.

Test Arm: Participants will either undergo Laparoscopic Sleeve Gastrectomy or Laparoscopic Gastric Bypass surgery. Approximately 9-13 months post bariatric surgery, each test arm participant will be evaluated to determine if he/she is still a candidate or if the need for knee replacement no longer exists (or is delayed). If the participant is still a candidate, he/she will undergo TKA. Participants will complete nine (9) research visits over the course of 3.5 - 4 years, in addition to the standard of care visits required for bariatric surgery and TKA. Research visits will include study activities such as vital sign measurements, orthopedic outcome assessments, physical function assessments (i.e. stair climb, 400 meter walk, etc.), questionnaire completion, and synovial fluid collection if the patient has a TKA procedure performed.

Control Arm: Participants in the control arm undergo a total knee replacement without surgical weight loss intervention and will complete six (6) research visits over the course of 2.5-3 years, in addition to the standard of care visits required for TKA. Research visits will include study activities such as vital sign measurements, orthopedic outcome assessments, physical function assessments (i.e. stair climb, 400 meter walk, etc.), questionnaire completion, and synovial fluid collection at the time of TKA.

The study hypothesis is that weight loss induced by bariatric surgery prior to TKA will improve TKA outcomes in patients with extreme obesity. The study hypothesis will be met if one of the following outcomes is achieved:

* In >=20% of bariatric surgery patients, the need for TKA was negated or delayed for at least two years.
* A statistically significant superiority is found among those patients undergoing bariatric surgery + TKA versus those undergoing TKA only in at least two of the following domains at two years post TKA:

  * Mobility (400 meter walk test)
  * Osteoarthritis outcome (WOMAC total score)
  * Knee orthopedic outcome (Knee Society score)
  * Quality of life (PROMIS-29 Quality of Life Questionnaire)
  * Osteoarthritic Pain (KOOS Pain)
  * Patient Satisfaction (If you had to live the rest of your life with the symptoms you have now, how would you feel?)

ELIGIBILITY:
Inclusion Criteria:

* Age 22-75 years.
* Subject is diagnosed with Non-inflammatory Degenerative Joint Disease(NIDJD).
* Subject is diagnosed with Morbid Obesity (Body Mass Index ≥ 40 kg/m2 or >35 kg/m2 with qualifying comorbid conditions such as obstructive sleep apnea or diabetes).
* Subject is a suitable candidate for cemented primary TKA with either resurfaced or non-resurfaced patellae.
* Subject is currently not bedridden.
* Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and co-operate with investigational procedures.
* Subject has given voluntary, written informed consent to participate in this clinical investigation.
* Subject is comfortable with speaking, reading, and understanding questions and providing responses in an available translated language.

Exclusion Criteria:

* Subject has undergone THA or contralateral knee within the past 6 months.
* Subject has had a contralateral amputation.
* Subject requires simultaneous bilateral TKA.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently experiencing radicular pain from the spine.
* Subject was diagnosed with fibromyalgia that is currently being treated with prescription medication.
* Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject has had previous bariatric surgery.
* Subject is medically or psychologically not suitable to undergo surgery.
* Subject is a known drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires.
* Subject has a medical condition with less than 2 years of life expectancy.
* Subject has participated in an IDE/IND clinical investigation with an investigational product in the last three months.
* Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is defined using the inclusion and exclusion criteria below. Demographic information (with the exclusion of age) is not used to determine the study population.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2016-01; Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of bariatric surgery patients who delay or no longer need TKA. | 1 year post bariatric surgery
  Participants in the Test Arm will undergo bariatric surgery prior to TKA. Determine if >=20% of Test Arm participants no longer need or delay the need for TKA.

SECONDARY OUTCOMES:
Mobility assessment using the 400 Meter Walk test | 2 years post TKA surgery
  Participants will be asked to complete 10 laps around cones that are 20 meters apart. During the test, participants will be asked to rate how hard they are walking and their level of knee pain. Heart rate and blood pressure will also be monitored. Mobility will be documented and analyzed to determine if there are changes throughout the course of the study.
Pain, disability and joint stiffness will be assessed using the Osteoarthritis Outcomes Questionnaire (WOMAC total score) | 2 years post TKA surgery
  The questionnaire is designed to assess pain, disability and joint stiffness in the osteoarthritis patient. Questionnaire answers will be documented and analyzed to determine if there are changes in pain, disability, and/or stiffness throughout the course of the study.
Pain, function, range of motion and joint stability will be assessed using the American Knee Society Score. | 2 years post TKA surgery
  The American Knee Society Score is an assessment and questionnaire that provides a rating of the pain, function, range of motion, and knee joint stability. It is subdivided into a knee score that rates only the knee joint itself and a functional score that rates the patient's ability to walk and climb stairs. Pain, function, range of motion, and joint stability will be documented and analyzed to determine if there are changes throughout the course of the study.
Quality of life will be assessed using the PROMIS-29 Quality of Life Questionnaire. | 2 years post TKA surgery
  Participants will be asked to complete a validated questionnaire known as PROMIS-29 to determine their quality of life. Answers to this questionnaire will be documented and analyzed to determine if there are changes in quality of life throughout the course of this study.
Knee pain will be assessed using the Osteoarthritic Pain Questionnaire (KOOS) | 2 years post TKA surgery
  The KOOS or Knee injury and Osteoarthritis Outcome Score are patient completed questionnaires which assess the patient's opinion regarding their knee and its associated osteoarthritis. Answers to this questionnaire will be documented and analyzed to determine if there are changes in knee pain throughout the course of this study.
Change in Patient Satisfaction | 2 years post TKA surgery
  Participants will be asked to answer the following question: If you had to live the rest of your life with the symptoms you have now, how would you feel? Answers to this question will be documented and analyzed to determine if there are changes in patient satisfaction throughout the course of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Still, DO, FACN, FACP, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Benotti P, Wood GC, Still C, Petrick A, Strodel W. Obesity disease burden and surgical risk. Surg Obes Relat Dis. 2006 Nov-Dec;2(6):600-6. doi: 10.1016/j.soard.2006.08.004. Epub 2006 Sep 22. PMID 16996319
- [Background] Friedman RJ, Hess S, Berkowitz SD, Homering M. Complication rates after hip or knee arthroplasty in morbidly obese patients. Clin Orthop Relat Res. 2013 Oct;471(10):3358-66. doi: 10.1007/s11999-013-3049-9. Epub 2013 May 14. PMID 23670675
- [Background] Malinzak RA, Ritter MA, Berend ME, Meding JB, Olberding EM, Davis KE. Morbidly obese, diabetic, younger, and unilateral joint arthroplasty patients have elevated total joint arthroplasty infection rates. J Arthroplasty. 2009 Sep;24(6 Suppl):84-8. doi: 10.1016/j.arth.2009.05.016. Epub 2009 Jul 15. PMID 19604665
- [Background] Namba RS, Paxton L, Fithian DC, Stone ML. Obesity and perioperative morbidity in total hip and total knee arthroplasty patients. J Arthroplasty. 2005 Oct;20(7 Suppl 3):46-50. doi: 10.1016/j.arth.2005.04.023. PMID 16214002
- [Background] Kerkhoffs GM, Servien E, Dunn W, Dahm D, Bramer JA, Haverkamp D. The influence of obesity on the complication rate and outcome of total knee arthroplasty: a meta-analysis and systematic literature review. J Bone Joint Surg Am. 2012 Oct 17;94(20):1839-44. doi: 10.2106/JBJS.K.00820. PMID 23079875
- [Background] Lozano LM, Nunez M, Segur JM, Macule F, Sastre S, Nunez E, Suso S. Relationship between knee anthropometry and surgical time in total knee arthroplasty in severely and morbidly obese patients: a new prognostic index of surgical difficulty. Obes Surg. 2008 Sep;18(9):1149-53. doi: 10.1007/s11695-008-9481-3. Epub 2008 May 28. PMID 18506553
- [Background] Severson EP, Singh JA, Browne JA, Trousdale RT, Sarr MG, Lewallen DG. Total knee arthroplasty in morbidly obese patients treated with bariatric surgery: a comparative study. J Arthroplasty. 2012 Oct;27(9):1696-700. doi: 10.1016/j.arth.2012.03.005. Epub 2012 May 2. PMID 22554730
- [Background] Kulkarni A, Jameson SS, James P, Woodcock S, Muller S, Reed MR. Does bariatric surgery prior to lower limb joint replacement reduce complications? Surgeon. 2011 Feb;9(1):18-21. doi: 10.1016/j.surge.2010.08.004. Epub 2010 Sep 27. PMID 21195326
- [Background] Parvizi J, Trousdale RT, Sarr MG. Total joint arthroplasty in patients surgically treated for morbid obesity. J Arthroplasty. 2000 Dec;15(8):1003-8. doi: 10.1054/arth.2000.9054. PMID 11112195
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] King WC, Engel SG, Elder KA, Chapman WH, Eid GM, Wolfe BM, Belle SH. Walking capacity of bariatric surgery candidates. Surg Obes Relat Dis. 2012 Jan-Feb;8(1):48-59. doi: 10.1016/j.soard.2011.07.003. Epub 2011 Jul 23. PMID 21937285
- [Background] Messier SP, Callahan LF, Golightly YM, Keefe FJ. OARSI Clinical Trials Recommendations: Design and conduct of clinical trials of lifestyle diet and exercise interventions for osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):787-97. doi: 10.1016/j.joca.2015.03.008. PMID 25952349
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Working Group on Health Outcomes for Older Persons with Multiple Chronic Conditions. Universal health outcome measures for older persons with multiple chronic conditions. J Am Geriatr Soc. 2012 Dec;60(12):2333-41. doi: 10.1111/j.1532-5415.2012.04240.x. Epub 2012 Nov 29. PMID 23194184
- [Background] Craig BM, Reeve BB, Brown PM, Cella D, Hays RD, Lipscomb J, Simon Pickard A, Revicki DA. US valuation of health outcomes measured using the PROMIS-29. Value Health. 2014 Dec;17(8):846-53. doi: 10.1016/j.jval.2014.09.005. PMID 25498780
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852